CLINICAL TRIAL: NCT01901302
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of CB-5945 for the Treatment of Opioid-Induced Constipation in Adults Taking Opioid Therapy for Chronic Non-Cancer Pain
Brief Title: Efficacy and Safety Study of CB-5945 for the Treatment of Opioid-Induced Constipation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision due to lack of enrollment.
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2402-003; 5945-OIC-12-02 (Other: Cubist Study Number)
Record Dates: First submitted 2013-07-09; First posted 2013-07-17 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Opioid-Induced Constipation
Keywords: Opioid; Constipation; Chronic; Pain
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CB-5945 (Experimental): 0.25 milligrams (mg) CB-5945 administered orally twice daily (BID) for a 12-week treatment period
  Interventions: Drug: CB-5945
- Placebo (Placebo Comparator): Placebo BID for a 12-week treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CB-5945
  Other Names: Bevenopran; ADL5945
  Arms: CB-5945
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CB-5945 for the treatment of opioid-induced constipation (OIC) in adults taking opioid therapy for chronic non-cancer pain.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, placebo-controlled, parallel-group study in participants with OIC taking opioid therapy for chronic non-cancer pain. Approximately 600 participants (300 participants per treatment group) with OIC will be randomized at approximately 75 study centers to receive either oral 0.25 mg CB-5945 BID or oral matching placebo BID for the 12-week double-blind treatment period, followed by a 4-week follow-up period. All randomized participants will be evaluated for clinical response for duration of their study participation. All participants will be followed for safety for 4 weeks after last dose of the study medication, regardless of when they discontinue study medication. The clinical study report for this study includes pooled results for studies 5945-OIC-12-02 (NCT01901302) 5945-OIC-12-03 (NCT01901328), and 5945-OIC-12-04 (NCT01901341).

ELIGIBILITY:
Key Inclusion Criteria:

* Is taking a stable daily dose of opioids of ≥30 mg morphine equivalent total daily dose (METDD) for chronic non-cancer pain
* Has constipation that is caused by the chronic use of opioids
* Is willing to use only the study provided laxative(s) and to discontinue use of all other laxatives, enemas, stool softeners, and other medications to treat constipation (e.g., lubiprostone) from Screening until the last study assessment

Key Exclusion Criteria:

* Has gastrointestinal (GI) or pelvic disorders known to affect bowel transit (for example [e.g.], obstruction) or contribute to bowel dysfunction
* Has evidence of intestinal obstruction
* Has a history of rectal bleeding not due to hemorrhoids or fissures within 6 months of screening
* Has an active malignancy of any type (participants with a history of successfully treated malignancy >5 years before the scheduled administration of study medication and participants with treated basal or squamous cell cancer may be enrolled)
* Is taking antispasmodics (e.g., dicyclomine), antidiarrheals (e.g., loperamide), prokinetics (e.g., metoclopramide), or locally acting chloride channel activators (e.g., lubiprostone)
* Is taking non-opioid medications known to cause constipation (e.g., iron sulfate therapy, tricyclic antidepressants)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-05-20 (Actual); Primary Completion 2014-02-13 (Actual); Study Completion 2014-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to difficulties with enrollment, this study was terminated early.
Groups:
- Placebo: Placebo administered orally BID for a 12-week treatment period
Period: Overall Study
Arm/Group | CB-5945 | Placebo
Started | 31 | 30
Received at Least 1 Dose of Study Drug | 31 | 30
Completed | 4 | 7
Not Completed | 27 | 23
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Study Terminated by Sponsor | 23 | 20
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomized to treatment who received ≥ 1 dose of double-blind study medication.
Groups:
- CB-5945: 0.25 mg CB-5945 administered orally BID for a 12-week treatment period
- Total: Total of all reporting groups
Arm/Group | CB-5945 | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 0 | 0
  BTWN | 31 | 27 | 58
  GTE65 | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Spontaneous Bowel Movement (SBM) Responder Rates at 12 Weeks
Description: A Spontaneous Bowel Movement (SBM) Weekly Responder (calculated for each week of the 12-week double-blind treatment period) is a participant who has ≥ 3 SBMs for the week and an increase from baseline of ≥1 SBM for the specified week, based on at least 4 Available Data Days (ADDs) during the week. A Complete SBM (CSBM) Weekly Responder is a participant who has ≥ 3 CSBMs for the specified week and an increase from baseline of ≥1 CSBM for the week.
  For the definition of the primary efficacy endpoint, Overall SBM Responder is a participant who is a Weekly SBM Responder for 9 of the 12 weeks of the double-blind treatment period, including 3 of the last 4 weeks (Weeks 9, 10, 11 and 12).
Time Frame: 12 weeks
Population: Zero participants were analyzed, and no data was collected for this measure. Due to lack of enrollment, the study was terminated early.
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline of Chronic Opioid-Related Gastrointestinal Symptom Scale (CORGISS) Scores at 12 Weeks
Description: The CORGISS is designed to assess GI symptoms related to opioid use in patients with chronic non-cancer pain. The CORGISS asks participants to rate the severity of GI symptoms over the previous 24 hours, with answers ranging from 0 ("did not experience") to 4 ("very severe").
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Complete Spontaneous Bowel Movement (CSBM) Responder Rates at 12 Weeks
Description: A CSBM Weekly Responder is a participant who has ≥ 3 CSBMs for the specified week and an increase from baseline of ≥1 CSBM for the week. An Overall CSBM Responder is a subject who is a Weekly CSBM Responder for 9 of the 12 weeks of the double-blind treatment period, including 3 of the last 4 weeks (Weeks 9, 10, 11 and 12).
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Adjudicated Cardiovascular, Gastrointestinal and Central Opioid Withdrawal Events
Description: Cardiovascular (CV) events of interested included mycardial infarction, unstable angina, cardiovascular accident, congestive heart failure, serious arrhythmia, resuscitated cardiac arrest, and death.
  Gastrointestinal (GI) events of interest included emergency department visits for SAEs of gastroenteritis, hepatitis, pancreatitis, nausea, vomiting, diarrhea, and abdominal pain or cramping.
  Central opioid withdrawal events of interest included opioid withdrawal syndrome.
Time Frame: Baseline through 16 weeks
Population: All participants randomized to treatment who received ≥ 1 dose of double-blind study medication.
Measure: Number; unit: participants
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 31 | 30
participants
  Subjects with at Least One Confirmed CV Event | 0 | 0
  Subjects with at Least One Confirmed GI Event | 0 | 0
  Subjects with at Least One Confirmed OW Event | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through 16 weeks
Arm/Group | CB-5945 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 9/31 | 8/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-5945 (N=31) | Placebo (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to difficulties with enrollment, this study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other